CLINICAL TRIAL: NCT07227519
Title: Online Randomized Experiment Evaluating Ultra-Processed Food Warning Labels on Social Media Posts Among Teens and Young Adults
Brief Title: Effects of UPF Warning Labels on Social Media Among Teens and Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Yuru Huang, Assistant Professor, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-10909-NHSR
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Nutrition; Healthy Diet; Food Preferences
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPF Warning Labels (Experimental): UPF warning labels will be placed beneath each social media post. Each label will feature an icon accompanied by explanatory text, using the exact health risk wording proposed in the Childhood Diabetes Reductions Act: "Warning: consuming ultra-processed foods and drinks can cause weight gain, which increases the risk of obesity and type-2 diabetes". All text will be left-aligned. The icon will consist of exclamation marks within a yellow triangle. The warning label will be large and highly visible and enclosed within a bold rectangular border.
  Interventions: Behavioral: UPF Warning Labels
- No Label (Control) (Other): No label
  Interventions: Behavioral: No Labels (Control)

INTERVENTIONS:
Behavioral: UPF Warning Labels — Participants will view four Instagram posts featuring UPFs, displayed with warning labels
  Arms: UPF Warning Labels
Behavioral: No Labels (Control) — Participants will view four Instagram posts featuring UPFs, displayed without warning labels
  Arms: No Label (Control)

SUMMARY:
This study aims to evaluate whether Ultra-Processed Food (UPF) warning labels on social media posts improve consumer understanding and influence purchase intentions among teens and young adults. Participants aged 13-29 in the United States will be recruited and randomized into two groups: a control group (no label) and an intervention group (UPF warning). Participants will view social media posts featuring UPFs with or without warning labels and respond to survey questions following each post.

DETAILED DESCRIPTION:
This study is designed to assess the effect of a highly visible UPF warning label on social media posts among adolescents and young adults in the United States. we will recruit approximately 500 US teens aged 13-17 and 500 young adults aged 18-29.

Participants will complete a between-subjects online randomized experiment. They will be randomized into either a UPF warning label group or a no label control group. Participants will view four social media posts featuring UPFs (with or without warning labels based on their assigned group) in random order. These posts are based on real Instagram advertisements from leading food and beverage companies; two posts will feature sugar-sweetened beverages and two will feature fast-food menu items. After viewing each post, participants will answer questions assessing consumer understanding, purchase intentions, and perceived healthfulness. At the end of the survey, all participants will also respond to questions regarding perceptions of control over healthy eating, policy support for UPF warnings, and their understanding of the term "ultra-processed food."

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-29
* Reside in the US
* Can read and speak English

Exclusion Criteria:

* Under the age of 13 or over 29
* Reside outside of the United States
* Unable to complete a survey in English

Ages: 13 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Consumer understanding | Assessed during one-time 10-minute online study survey
  For each social media post, participants will be asked whether they think the product is ultra-processed. Response options will be "yes", "no", or "I don't know". Consumer understanding will be coded as a binary outcome: "yes" = correct; "no" and "I don't know" = incorrect.
Purchase intentions | Assessed during one-time 10-minute online study survey
  For each social media post, participants will be asked how likely they would buy the product in the next week, either in-store or online. Response options will be on a 1-5 Likert scale, with 5 being "very likely". Higher scores indicate higher intentions to purchase the product.

SECONDARY OUTCOMES:
Perceived healthfulness | Assessed during one-time 10-minute online study survey
  For each social media post, participants will be asked how healthy the product seems to them. Responses options will be on a 1-5 Likert scale, with 5 indicating "very healthy". Higher scores indicate higher perceived healthfulness.
Perceptions of control over healthy eating | Assessed during one-time 10-minute online study survey
  After viewing all four social media posts, all participants will be shown the UPF warning label (regardless of condition) and asked whether the UPF warning labels make them feel "less in control of making healthy eating decision," "neither less nor more in control or making healthy eating decisions," or "more in control of making healthy eating decisions." Responses will be binary coded: "more in control" = 1; "less" or "neither" = 0.
Policy support for ultra-processed food warning labels | Assessed during one-time 10-minute online study survey
  After viewing all four social media posts, all participants will be shown the UPF warning label (regardless of condition) and asked whether they support or oppose a policy requiring these labels on social media advertisements for ultra-processed foods and beverages. Response options will be on a 1-5 Likert scale, with 5 indicating "Strongly support." Higher scores will indicate higher support for warning labels.

CONTACTS AND LOCATIONS:
Overall Officials: Yuru Huang, Principal Investigator — University of Tennessee; Anna Grummon, Principal Investigator — Stanford University
Locations (1):
- UTHSC Department of Preventive Medicine, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will post de-identified individual participant data in a public repository.
Supporting Information: SAP, Analytic Code
Time Frame: Investigators will post IDP within 6 months of publication of manuscripts associated with the data generated in this study.
Access Criteria: Data and code will be made publicly available.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT07227519/SAP_002.pdf